CLINICAL TRIAL: NCT07206498
Title: A Phase I/II Study to Evaluate Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of WSD0922-FU in Combination With Osimertinib for Patients With Locally Advanced or Metastatic Non- Small Cell Lung Cancer
Brief Title: A Study to Evaluate Safety and Efficacy of WSD0922-FU Combo With Osimertinib for NSCLC
Acronym: WAYWIN103
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayshine Biopharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WSD0922-103
Record Dates: First submitted 2025-09-19; First posted 2025-10-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: WSD0922; WSD0922-FU; NSCLC; CNS metastasis; Brain metastasis; EGFR; C797S; Del19; L858R
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Part A (Dose escalation study) ; Part B (Does expansion study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation (WSD0922-FU and Osimertinib) (Experimental): Patients receive 80mg Osimertinib PO QD and WSD0922-FU PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and blood sample collection on study.
  Interventions: Drug: Osimertinib (Tagrisso®); Drug: WSD0922-FU
- Dose expansion (WSD0922-FU and Osimertinib) (Experimental): Patients receive 80mg Osimertinib PO QD and WSD0922-FU PO QD using dosage selected from Dose escalation. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and blood sample collection on study.
  Interventions: Drug: Osimertinib (Tagrisso®); Drug: WSD0922-FU

INTERVENTIONS:
Drug: Osimertinib (Tagrisso®) — Drug: Osimertinib Procedure: Biospecimen Collection - blood samples Undergo collection of blood samples
  Procedure: Computed Tomography and/or Magnetic Resonance Imaging Undergo CT and/or MRI
  Drug: Osimertinib Given PO, 80mg, once daily
Drug: WSD0922-FU — Drug: WSD0922-FU Procedure: Biospecimen Collection - blood samples Undergo collection of blood samples
  Procedure: Computed Tomography and/or Magnetic Resonance Imaging Undergo CT and/or MRI
  Drug: WSD0922-FU Given PO

SUMMARY:
This is a Phase I/II, Open Label Study of WSD0922-FU in Combination with Osimertinib for Patients with Locally Advanced or Metastatic Non-Small Cell Lung Cancer whose disease has progressed with third-generation EGFR-TKI with C797S mutation or is newly diagnosed with CNS metastasis with EGFR Del19 or L858R mutation

DETAILED DESCRIPTION:
WSD0922-FU is a potent reversible inhibitor of both the single EGFRm+ and dual EGFRm+/C797S+ receptor forms of EGFR with selectivity margin over wild-type EGFR. This study aims to explore the safety, tolerability, pharmacokinetic characteristics and efficacy of WSD0922-FU combined with Osimertinib in patients with non-small cell lung cancer (NSCLC) with C797S mutation after first-line third-generation EGFR-TKI resistance, and then further confirm the safety and efficacy for newly diagnosed NSCLC BM patients with classical EGFR Del19 or L858R mutation

ELIGIBILITY:
Inclusion Criteria:

* ≥Age 18, gender is not limited;
* Locally advanced or metastatic NSCLC confirmed by pathology;
* Patients who have been genetically tested to carry EGFR sensitive mutations;
* Blood/Tissue samples must be provided for testing;
* Must have a minimum life expectancy of >= 3 months;
* At least one measurable tumor lesion according to RECIST version 1.1; ● Previous radiotherapy-treated lesions cannot be used as target lesions unless imaging studies show clear progression of the lesions.
* Physical Status (ECOG PS) score was 0-1;
* Have full organ function;
* Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method ;
* Subjects are required to give informed consent to this study before the experiment and sign a written informed consent voluntarily.

Exclusion Criteria:

* Received chemotherapy, radiotherapy, biological therapy, targeted therapy, endocrine therapy, immunotherapy, or other anti-tumor drug treatments within 4 weeks before the first administration of the study drug.
* Have previously received more than two EGFR-TKI inhibitors for part A;
* Received major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks before the first administration, or require elective surgery during the trial period.
* Used strong CYP3A4 inhibitors or strong CYP3A4 inducers within 7 days before the first use of the study drugs.
* Adverse reactions from previous anti-tumor treatments have not recovered to NCI-CTCAE v5.0 grade ≤1 (except for toxicities judged by the researcher to have no safety risks, such as hair loss, grade 2 peripheral neurotoxicity, and stable thyroid function after hormone replacement therapy).
* Skin/pressure ulcers, chronic leg ulcers, known active gastric ulcers, or non-healing wounds.
* History of severe allergies, or allergies to any active or inactive ingredients of the study drug;
* Severe infections requiring intravenous antibiotic infusion or hospitalization at the time of screening; or uncontrollable active infections within 4 weeks before administration;
* Known active or suspected autoimmune diseases; or known active ocular diseases (such as active wet age-related macular degeneration, diabetic retinopathy with macular edema);
* Human immunodeficiency virus (HIV) (HIV1/2 antibody) positive, syphilis spirochete antibody positive .
* Patients with interstitial lung disease.
* History of severe cardiovascular diseases.
* Unable to orally swallow medication, or there is a condition that significantly affects gastrointestinal absorption as judged by the researcher; Clinical intervention is required for pleural effusion, ascites (excluding subjects who do not need drainage and have been stable for more than 2 weeks after drainage).
* Known alcohol or drug dependence.
* Mental disorders or poor compliance;
* Pregnant or lactating women;
* The investigator believes that the subject has other reasons that make them unsuitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-10-14 (Estimated); Study Completion 2029-10-14 (Estimated)

PRIMARY OUTCOMES:
PartA: To evaluate the safety of WSD0922-FU combined with Osimertinib in patients with NSCLC | 12 months
  Safety (incidence and severity of adverse events [AE])
PartB: To evaluate the efficacy of WSD0922-FU combined with Osimertinib in patients with NSCLC | every 6 weeks, up to 2 years
  ORR

SECONDARY OUTCOMES:
To evaluate the safety of WSD0922-FU in patients with advanced non-small cell lung cancer | 12 months
  Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Adverse Events (TRAEs)
Disease Control Rate (DCR) | every 6 weeks, up to 24 months
  the percentage of patients who have a best overall response of CR or PR or SD
Duration of Response (DoR) | every 6 weeks, up to 24 months
  proportion of patients with the time from the date of first documented response until the date of documented progression or death in the absence of disease progression
PFS | every 6 weeks, up to 24 months
  proportion of patients with the time from randomization until the date of objective disease progression or death
Intracranial Disease Control Rate (iDCR) | every 6 weeks, up to24 months
  the percentage of patients who have a best overall response of CR or PR or SD per RANO BM
Intracranial Duration of Response (iDoR) | every 6 weeks, up to 24 months
  proportion of patients with the time from the date of first documented response until the date of documented progression or death in the absence of disease progression per RANO BM
iPFS | every 6 weeks, up to 24 months
  proportion of patients with the time from randomization until the date of objective disease progression or death per RANO BM

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No